CLINICAL TRIAL: NCT01273454
Title: An Open-label, Multi-center, Non-interventional Study to Investigate Clinical Usefulness of Hydromorphone OROS in Korean Cancer Patients
Brief Title: An Observational Study to Investigate Clinical Usefulness of OROS Hydromorphone in Korean Cancer Patients
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016324
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Pain
Keywords: Open-label; Non-interventional; OROS hydromorphone; Korean cancer patients
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001: OROS Hydromorphone 8 16 32 mg once a day for 4 weeks
  Interventions: Drug: OROS Hydromorphone

INTERVENTIONS:
Drug: OROS Hydromorphone — 8,16, 32 mg once a day for 4 weeks

SUMMARY:
This study aims to collect clinical information and to examine the usefulness and safety of ORal Osmotic System Hydromorphone in Korean cancer patients. The decision to treat patients with drug is as per physician discretion and that doses are determined based upon approved labeling recommendations and physician discretion.

DETAILED DESCRIPTION:
The primary purpose of this observational study is to collect clinical data on cancer pain control using OROS (ORal Osmotic Active System) hydromorphone and to investigate the clinical usefulness of OROS hydromorphone for Korean cancer patients. Information on the effectiveness of cancer pain control and any adverse events reported by those patients using OROS Hydromorphone will be reported. In addition, clinical usefulness of OROS hydromorphone will be evaluated through assessing sleep disturbance due to pain, breakthrough pain, and end-of-dose failure before and after the study drug administration and examining the patient's satisfaction with study drug and the investigator's global assessment. This is a multi-center, open-label, prospective, exploratory, and observational study with approximately 770 patients. Efficacy endpoints will be analyzed to examine the difference between before and after the treatment. Since this is an observational study under the condition of routine practice, OROS Hydromorphone dosage should be adjusted at the discretion of the investigator, based on patient response. It is recommended that the dosage be conservative at first and adjusted appropriately considering the adverse events and analgesic effect for all the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are in need OROS hydromorphone to relieve cancer pain

Exclusion Criteria:

* Patients with serious gastrointestinal diseases that may interfere with oral analgesic effects, such as dysphagia, vomiting, absence of periastalsis, intestinal obstruction, and/or severe strangulation, in which case the absorption and passage of orally-administered medication may be unduly influenced

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from cancer pain who visit the study sites during study and eligible to be treated with OROS hydromorphone at the discretion of the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 648 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity score (where 0 is worst and 10 is best) as measured on the Numeric Rating Scale (NRS) from baseline to Day 36 | Between Visit 1 (day 1) and the last visit (day 29 ± 7: from day 22 to day 36)

SECONDARY OUTCOMES:
Change in sleep disturbance | between Visit 1 (DAY 1) and the last visit (DAY29 ± 7: from 22 day to 36 day))
Breakthrough pain experience | between Visit 1 (DAY 1) and the last visit (DAY29 ± 7: from 22 day to 36 day))
End-of-dose failure experience | between Visit 1 (DAY 1) and the last visit (DAY29 ± 7: from 22 day to 36 day))
Patient satisfaction with study drug and detailed reason | at the last visit (DAY29 ± 7: from 22 day to 36 day))
Investigator's global assessment | the last visit (DAY29 ± 7: from 22 day to 36 day)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

REFERENCES:
- [Derived] Park CK, Kang HW, Oh IJ, Kim YC, Kim YK, Na KJ, Ahn SJ, Kim TO, Choi YJ, Song GA, Lee MK. Once-Daily OROS Hydromorphone for Management of Cancer Pain: an Open-Label, Multi-Center, Non-Interventional Study. J Korean Med Sci. 2016 Dec;31(12):1914-1921. doi: 10.3346/jkms.2016.31.12.1914. PMID 27822929